CLINICAL TRIAL: NCT04896658
Title: Belantamab Mafodotin, Cyclophosphamide and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Brief Title: Belantamab Mafodotin, Cyclophosphamide, and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to FDA withdrawal of the drug and lack of enrollment with available BCMA therapies that were deemed safer.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ashraf Badros, Director of Multiple Myeloma Service, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2060GCCC
Record Dates: First submitted 2021-01-13; First posted 2021-05-21 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Belantamab mafodotin; Relapsed/Refractory Multiple Myeloma; Maximum tolerated doses; Overall response rate; Overall survival; Dose limiting toxicities
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase I
  1. Arm A (cycles repeated every 3 weeks)
     1. Dose level 1: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
     2. Dose level 2: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
  2. Arm B (cycles repeated every 6 weeks)
     1. Dose level 1: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
     2. Dose level 2: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
  Phase II : Phase II was stopped with the FDA withdrawal of the drug approval and reluctance of patients to participate.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): 1. Dose level 1: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
  2. Dose level 2: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 3 weeks cycles.
  Interventions: Drug: Belantamab Mafodotin, Cyclophosphamide and Dexamethasone
- Arm B (Experimental): 1. Dose level 1: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
  2. Dose level 2: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 6 weeks cycles.
  Interventions: Drug: Belantamab Mafodotin, Cyclophosphamide and Dexamethasone

INTERVENTIONS:
Drug: Belantamab Mafodotin, Cyclophosphamide and Dexamethasone — Study drug

SUMMARY:
Evaluate the efficacy and safety of Belantamab Mafodotin, cyclophosphamide, and dexamethasone in patients with Relapsed/Refractory Multiple Myeloma

DETAILED DESCRIPTION:
This is a Phase I/II, open-label study to evaluate the efficacy and safety of Belantamab Mafodotin, cyclophosphamide, and dexamethasone.

In Phase I, the subjects will be assigned into two arms and there are two dose levels for Belantamab Mafodotin and there are two dose levels of cyclophosphamide in each arm.

In Phase II, once tolerability of the highest planned dose is established, the patients will be assessed for response rate. The arm with acceptable toxicity and best response will be further assessed in the expansion cohort.

Belantamab mafodotin was approved by the U.S. Food and Drug Administration (FDA) on Aug 5, 2020, for treating patients with relapsed/refractory multiple myeloma. Cyclophosphamide and dexamethasone are both approved by the FDA. But the combinations with these three drugs to treat people with relapsed/refractory multiple myeloma has not been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of Refractory MM; failed at least 3 prior lines of anti-myeloma treatments, including an anti-CD38 antibody (e.g., daratumumab) alone or in combination, and is refractory to an IMiD (i.e., lenalidomide or pomalidomide), and to a proteasome inhibitor (e.g., bortezomib, ixazomib or carfilzomib). (Refractory myeloma is defined as disease that is nonresponsive while on primary or salvage therapy or progresses within 60 days of last therapy. Nonresponsive disease is defined as either failure to achieve at least minimal response or development of progressive disease (PD) while on therapy).
2. Has measurable disease with at least one of the following:

   1. Serum M-protein ≥0.5 g/dL (≥ 5 g/L)
   2. Urine M-protein ≥ 200 mg/24h
   3. Serum FLC assay: Involved FLC level ≥10 mg/dL and an abnormal ratio (<0.26 or >1.65)
3. Provide signed written informed consent.
4. 18 years or older (at the time consent is obtained).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Participants with a history of autologous stem cell transplant or Prior BCMA targeted therapy (e.g. CAR-T cells, BiTes) can enroll on the study provided that:

   1. Therapy was >100 days prior to study enrolment.
   2. No active infection(s).
7. Adequate organ system function (as defined by inclusion criteria #7).
8. Female and Male patients: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
9. Prior treatment-related toxicities must be ≤ Grade 1 except peripheral neuropathy (Grade-2).

Exclusion Criteria:

1. Systemic anti-myeloma therapy within ≤14 days or 5 half-lives, whichever is shorter, or plasmapheresis within 7 days prior to treatment.
2. Systemic treatment with high dose steroids (equivalent to ≥ 60 mg prednisone daily for ≥4 days) within the past 14 days.
3. Symptomatic amyloidosis, active CNS disease, active plasma cell leukemia at the time of screening.
4. Prior allogeneic stem cell transplant (SCT). NOTE - Participants who have undergone syngeneic transplant may be allowed if no history of GvHD.
5. Current corneal epithelial disease except mild punctate keratopathy.
6. Evidence of active bleeding.
7. Any major surgery within the last four weeks.
8. Presence of active renal condition (infection, dialysis); isolated proteinuria from MM is allowed provided participants fulfil the adequate organ system function criteria (as defined by inclusion criteria #7).
9. Any serious and/or unstable pre-existing medical, psychiatric disorder or lab abnormalities that affect patients' safety, obtaining informed consent or compliance with study procedures.
10. Current unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
11. Other malignancies except for malignancy from which the patients have been disease-free > 2 years.
12. Evidence of cardiovascular disease including any of the following:

    1. Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including second degree (Mobitz Type II) or third degree atrioventricular (AV) block.
    2. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening.
    3. Class III or IV heart failure as defined by the New York Heart Association functional classification system.
    4. Uncontrolled hypertension.
13. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, daratumumab, bortezomib, boron or mannitol or any other components of the study treatment.
14. Active infection requiring treatment.
15. Known HIV infection.
16. Presence of hepatitis B surface antigen (HbsAg), or hepatitis B core antibody (HbcAb), at screening or within 3 months prior to first dose of study treatment. Note: presence of Hep B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant.
17. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

    NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
18. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
19. Pregnant or lactating female.
20. Concomitant administration of strong P-glycoprotein inhibitors and inhibitors of OATP will be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Badros, MB; ChB, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alley SC, Zhang X, Okeley NM, Anderson M, Law CL, Senter PD, Benjamin DR. The pharmacologic basis for antibody-auristatin conjugate activity. J Pharmacol Exp Ther. 2009 Sep;330(3):932-8. doi: 10.1124/jpet.109.155549. Epub 2009 Jun 4. PMID 19498104
- [Background] Chari A, Vogl DT, Gavriatopoulou M, Nooka AK, Yee AJ, Huff CA, Moreau P, Dingli D, Cole C, Lonial S, Dimopoulos M, Stewart AK, Richter J, Vij R, Tuchman S, Raab MS, Weisel KC, Delforge M, Cornell RF, Kaminetzky D, Hoffman JE, Costa LJ, Parker TL, Levy M, Schreder M, Meuleman N, Frenzel L, Mohty M, Choquet S, Schiller G, Comenzo RL, Engelhardt M, Illmer T, Vlummens P, Doyen C, Facon T, Karlin L, Perrot A, Podar K, Kauffman MG, Shacham S, Li L, Tang S, Picklesimer C, Saint-Martin JR, Crochiere M, Chang H, Parekh S, Landesman Y, Shah J, Richardson PG, Jagannath S. Oral Selinexor-Dexamethasone for Triple-Class Refractory Multiple Myeloma. N Engl J Med. 2019 Aug 22;381(8):727-738. doi: 10.1056/NEJMoa1903455. PMID 31433920
- [Background] Dougherty BE, Nichols JJ, Nichols KK. Rasch analysis of the Ocular Surface Disease Index (OSDI). Invest Ophthalmol Vis Sci. 2011 Nov 7;52(12):8630-5. doi: 10.1167/iovs.11-8027. PMID 21948646
- [Background] Gandhi UH, Cornell RF, Lakshman A, Gahvari ZJ, McGehee E, Jagosky MH, Gupta R, Varnado W, Fiala MA, Chhabra S, Malek E, Mansour J, Paul B, Barnstead A, Kodali S, Neppalli A, Liedtke M, Narayana S, Godby KN, Kang Y, Kansagra A, Umyarova E, Scott EC, Hari P, Vij R, Usmani SZ, Callander NS, Kumar SK, Costa LJ. Outcomes of patients with multiple myeloma refractory to CD38-targeted monoclonal antibody therapy. Leukemia. 2019 Sep;33(9):2266-2275. doi: 10.1038/s41375-019-0435-7. Epub 2019 Mar 11. PMID 30858549
- [Background] Heylmann D, Bauer M, Becker H, van Gool S, Bacher N, Steinbrink K, Kaina B. Human CD4+CD25+ regulatory T cells are sensitive to low dose cyclophosphamide: implications for the immune response. PLoS One. 2013 Dec 23;8(12):e83384. doi: 10.1371/journal.pone.0083384. eCollection 2013. PMID 24376696
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Laurent SA, Hoffmann FS, Kuhn PH, Cheng Q, Chu Y, Schmidt-Supprian M, Hauck SM, Schuh E, Krumbholz M, Rubsamen H, Wanngren J, Khademi M, Olsson T, Alexander T, Hiepe F, Pfister HW, Weber F, Jenne D, Wekerle H, Hohlfeld R, Lichtenthaler SF, Meinl E. gamma-Secretase directly sheds the survival receptor BCMA from plasma cells. Nat Commun. 2015 Jun 11;6:7333. doi: 10.1038/ncomms8333. PMID 26065893
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] Macsai M, Nariani A, Gan H, Lassman A, Merrell R, Gomez E, et al. Corneal Toxicity of ABT-414 in Glioblastoma (GBM): Clinical Manifestations, Ophthalmological Findings and Management. Investigative Ophthalmology & Visual Science. 2016 Sep 26;57(12):269-269.
- [Background] Xie J, He Y. Ontology-Based Vaccine Adverse Event Representation and Analysis. Adv Exp Med Biol. 2017;1028:89-103. doi: 10.1007/978-981-10-6041-0_6. PMID 29058218
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Pirogova OV, Moiseev IS, Surkova EA, Lapin SV, Bondarenko SN, Kulagin AD, Afanasyev BV. Profiles of pro-inflammatory cytokines in allogenic stem cell transplantation with post-transplant cyclophosphamide. Cytokine. 2017 Nov;99:148-153. doi: 10.1016/j.cyto.2017.08.016. Epub 2017 Sep 9. PMID 28898706
- [Background] Roghanian A, Hu G, Fraser C, Singh M, Foxall RB, Meyer MJ, Lees E, Huet H, Glennie MJ, Beers SA, Lim SH, Ashton-Key M, Thirdborough SM, Cragg MS, Chen J. Cyclophosphamide Enhances Cancer Antibody Immunotherapy in the Resistant Bone Marrow Niche by Modulating Macrophage FcgammaR Expression. Cancer Immunol Res. 2019 Nov;7(11):1876-1890. doi: 10.1158/2326-6066.CIR-18-0835. Epub 2019 Aug 26. PMID 31451483
- [Background] Sanchez E, Li M, Kitto A, Li J, Wang CS, Kirk DT, Yellin O, Nichols CM, Dreyer MP, Ahles CP, Robinson A, Madden E, Waterman GN, Swift RA, Bonavida B, Boccia R, Vescio RA, Crowley J, Chen H, Berenson JR. Serum B-cell maturation antigen is elevated in multiple myeloma and correlates with disease status and survival. Br J Haematol. 2012 Sep;158(6):727-38. doi: 10.1111/j.1365-2141.2012.09241.x. Epub 2012 Jul 18. PMID 22804669
- [Background] Tai YT, Li XF, Breitkreutz I, Song W, Neri P, Catley L, Podar K, Hideshima T, Chauhan D, Raje N, Schlossman R, Richardson P, Munshi NC, Anderson KC. Role of B-cell-activating factor in adhesion and growth of human multiple myeloma cells in the bone marrow microenvironment. Cancer Res. 2006 Jul 1;66(13):6675-82. doi: 10.1158/0008-5472.CAN-06-0190. PMID 16818641
- [Background] Thompson JA, Motzer RJ, Molina AM, Choueiri TK, Heath EI, Redman BG, Sangha RS, Ernst DS, Pili R, Kim SK, Reyno L, Wiseman A, Trave F, Anand B, Morrison K, Donate F, Kollmannsberger CK. Phase I Trials of Anti-ENPP3 Antibody-Drug Conjugates in Advanced Refractory Renal Cell Carcinomas. Clin Cancer Res. 2018 Sep 15;24(18):4399-4406. doi: 10.1158/1078-0432.CCR-18-0481. Epub 2018 May 30. PMID 29848572
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Anderson LD Jr, Sutherland HJ, Yong K, Hoos A, Gorczyca MM, Lahiri S, He Z, Austin DJ, Opalinska JB, Cohen AD. Targeting B-cell maturation antigen with GSK2857916 antibody-drug conjugate in relapsed or refractory multiple myeloma (BMA117159): a dose escalation and expansion phase 1 trial. Lancet Oncol. 2018 Dec;19(12):1641-1653. doi: 10.1016/S1470-2045(18)30576-X. Epub 2018 Nov 12. PMID 30442502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: 12/03/2021- 01/08/2024 Types of location: UMGCCC outpatient clinic
Pre-assignment Details: Reasons for exclusion- history of GvHD; wears scleral lenses, Patient withdrew consent, No Measurable Disease, Inadequate organ system function, Current unstable liver disease
Groups:
- Phase I: Arm A: 1. Dose level 1: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
  2. Dose level 2: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 3 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Phase 1: Arm B: 1. Dose level 1: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
  2. Dose level 2: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 6 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
Period: Dose Level 1
Arm/Group | Phase I: Arm A | Phase 1: Arm B
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Dose Level 2
Arm/Group | Phase I: Arm A | Phase 1: Arm B
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total enrollment was 10. 3 patients were enrolled in Phase I: Arm A - Dose level 1. 3 participants were enrolled in Phase I Arm B - Dose level 1. 4 participants were enrolled in Phase I Arm B - Dose level 2.
Groups:
- Phase I: Arm A - Dose Level 1: (1) Dose level 1: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Phase I: Arm A - Dose Level 2: (2) Dose level 2: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 3 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Phase I: Arm B - Dose Level 1: (1) Dose level 1: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Phase I: Arm B - Dose Level 2: (2) Dose level 2: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 6 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Total: Total of all reporting groups
Arm/Group | Phase I: Arm A - Dose Level 1 | Phase I: Arm A - Dose Level 2 | Phase I: Arm B - Dose Level 1 | Phase I: Arm B - Dose Level 2 | Total
Number analyzed (Participants) | 3 | 0 | 3 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: Total enrollment was 10. 3 patients were enrolled in Part A and 7 participants were enrolled in Part B
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0 | 1 | 1
    >=65 years | 3 | 0 | 3 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 3 | 5
  Male | 2 | 0 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 1 | 0 | 3 | 2 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events in Dose Escalation
Description: Overall incidence and severity of Adverse Events in Number of Participants with Adverse Events in Dose Escalation
Time Frame: Up to 6 weeks
Population: 3 patients were enrolled in Arm A, Dose Level 1. Arm A was closed due to AEs and no patients enrolled in Arm A, Dose Level 2 3 patients were enrolled in Arm B, Dose Level 1. Then 4 new patients were enrolled in Arm B, Dose Level 2.
  Part 2 was stopped with the FDA withdrawal of the drug approval and reluctance of patients to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A - Dose Level 1: (1) Dose level 1: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 3 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Arm A - Dose Level 2: (2) Dose level 2: The subject will take 1.9 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 3 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Arm B - Dose Level 1: (1) Dose level 1: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 300 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 of each 6 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
- Arm B - Dose Level 2: (2) Dose level 2: The subject will take 2.5 mg/kg of Belantamab Mafodotin, 500 mg of Cyclophosphamide, and 40 mg of Dexamethasone on day 1 each 6 weeks cycles.
  Belantamab Mafodotin, Cyclophosphamide and Dexamethasone: Study drug
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm B - Dose Level 1 | Arm B - Dose Level 2
Number analyzed (Participants) | 3 | 0 | 3 | 4
Participants | 3 | 0 | 3 | 4

2. Primary Outcome: Response Rate in Dose Escalation and Expansion Cohort
Description: Number of Participants With response rate in Dose Escalation and Expansion Cohort. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 weeks
Population: Phase II of the expansion cohort was stopped with the FDA withdrawal of the drug approval and reluctance of patients to participate. 0 patients were enrolled in the Phase II expansion Cohort, therefore, there is no data to report in the data table.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II : Expansion Cohort: Once tolerability of the highest planned dose is established, patients will be assessed for response rate. The arm with acceptable toxicity and best response will be further assessed in the expansion cohort.
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Phase II : Expansion Cohort
Number analyzed (Participants) | 3 | 0 | 3 | 4 | 0
Participants | 3 | 0 | 3 | 4 | 0

3. Secondary Outcome: Number of Participants With Disease Progression
Description: Number of participants with disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of randomization until the date of death from any cause, assessed up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Phase II : Expansion Cohort
Number analyzed (Participants) | 3 | 0 | 3 | 4 | 0
Participants | 0 | 0 | 1 | 3 | 0

4. Secondary Outcome: Number of Participants According to Best Response
Description: Best Response (Not including Overall Survival (OS) response)
Time Frame: From date of randomization until the date of death from any cause, assessed up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Phase II : Expansion Cohort
Number analyzed (Participants) | 3 | 0 | 3 | 4 | 0
Participants
  Stable Disease (SD) | 1 | 0 | 2 | 2 | 0
  Partial Response (PR) | 2 | 0 | 1 | 1 | 0
  Very good partial response (VGPR) | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Overall Survival
Description: Number of patients with overall survival response
Time Frame: From date of randomization until the date of death from any cause, assessed up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Phase II : Expansion Cohort
Number analyzed (Participants) | 3 | 0 | 3 | 4 | 0
Participants | 2 | 0 | 3 | 3 | 0

6. Other Pre Specified Outcome: Cytokine Profile Data
Description: The cytokines were exploratory data, and were done on few patients, data is not conclusive to establish a reasonable ink with toxicity. Therefore, this endpoint cannot be provided.
Time Frame: From date of randomization until the date of death from any cause, assessed up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed through study completion, up to 3 years; all adverse events were collected through 6 weeks
Description: Arm A was stopped and 0 patients were enrolled in Arm A - Dose Level 2. Therefore, there were no participants at risk for Serious Adverse Events or for All-Cause Mortality in Arm A - Dose Level 2.
Arm/Group | Phase I: Arm A - Dose Level 1 | Phase I: Arm A - Dose Level 2 | Phase I: Arm B - Dose Level 1 | Phase I: Arm B - Dose Level 2
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/0 | 0/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 2/3 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Arm A - Dose Level 1 (N=3) | Phase I: Arm A - Dose Level 2 (N=0) | Phase I: Arm B - Dose Level 1 (N=3) | Phase I: Arm B - Dose Level 2 (N=4)
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Ablation (Cardiac disorders) | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — R distal dorsal forearm
Fracture, Right Humerus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Arm A - Dose Level 1 (N=3) | Phase I: Arm A - Dose Level 2 (N=0) | Phase I: Arm B - Dose Level 1 (N=3) | Phase I: Arm B - Dose Level 2 (N=4)
Abdominal Pain (General disorders) | 0 | 0 | 0 | 1
Acute cystitis without hematuria (Infections and infestations) | 0 | 0 | 0 | 1
Allergic Rhinitis (General disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anemia B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Blurred Vision (Eye disorders) | 3 | 0 | 1 | 1
Bilateral Epithelial Edema (General disorders) | 0 | 0 | 1 | 0
Bilateral hyperopic shift (Eye disorders) | 0 | 0 | 1 | 0
bilateral Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 1 | 0
Superficial punctate keratopathy (Eye disorders) | 2 | 0 | 1 | 0
Bilateral Subepithelial Haze (Eye disorders) | 0 | 0 | 1 | 0
Bilateral superficial epithelial microcyst-like changes (Eye disorders) | 2 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 1
Chin Neuropathy (General disorders) | 0 | 0 | 1 | 0
Chronic Epiretinal Membrane (right eye) (Eye disorders) | 0 | 0 | 1 | 0
Cold (General disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Back Pain (General disorders) | 1 | 0 | 0 | 1
Central Corneal cysts with overlying Punctate Epithelial Erosions [PEE] (Eye disorders) | 1 | 0 | 0 | 0
Cough (General disorders) | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
diffuse microcyst involving the central visual axis (Eye disorders) | 1 | 0 | 0 | 0
Dizziness (General disorders) | 0 | 0 | 1 | 0
Dry eyes (Eye disorders) | 0 | 0 | 0 | 1
Dry skin rash (General disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Facial neuropathy (General disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Corneal Changes (Eye disorders) | 3 | 0 | 2 | 1
Ocular Toxicity (Eye disorders) | 0 | 0 | 0 | 1
Gum pain (General disorders) | 0 | 0 | 0 | 1
Headaches (General disorders) | 1 | 0 | 0 | 1
Hiccups (General disorders) | 0 | 0 | 1 | 0
Hip and groin pain (General disorders) | 1 | 0 | 0 | 0
Humerus fracture, left (General disorders) | 0 | 0 | 0 | 1
Hypertension (General disorders) | 2 | 0 | 1 | 0
Hypocalcemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypokalemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
hypomagnesemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Imbalance sensation (General disorders) | 0 | 0 | 0 | 1
Increased bilirubin (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Intermittent Gastroesophageal Reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Leg Pain (General disorders) | 1 | 0 | 0 | 1
Muscle Cramps (General disorders) | 1 | 0 | 0 | 0
Nasal congestion (General disorders) | 0 | 0 | 1 | 0
Nausea (General disorders) | 0 | 0 | 0 | 2
Otitis externa (General disorders) | 1 | 0 | 0 | 0
Parainfluenza Virus (General disorders) | 0 | 0 | 0 | 1
Peripheral Corneal cysts with Mild Punctate Epithelial Erosions [PEE] (Eye disorders) | 1 | 0 | 0 | 0 — right eye
Peripheral sensory neuropathy (General disorders) | 0 | 0 | 0 | 1 — - left hand
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Postnasal drip (General disorders) | 0 | 0 | 1 | 0
Productive cough (General disorders) | 0 | 0 | 0 | 1
Rash (General disorders) | 1 | 0 | 0 | 0
Fracture (General disorders) | 0 | 0 | 0 | 1 — right arm
Hip pain (General disorders) | 0 | 0 | 0 | 1 — right hip
Lesion (General disorders) | 1 | 0 | 0 | 0 — right lower leg
Runny nose (General disorders) | 0 | 0 | 1 | 0
Scleral disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — burst blood vessel in right eye
Itchy eyes (Eye disorders) | 0 | 0 | 1 | 0
Sore throat (General disorders) | 0 | 0 | 1 | 1
Stomach Pain (General disorders) | 1 | 0 | 0 | 0
Upset Stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary Tract Infection (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Vitamin B6 deficiency (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04896658/Prot_SAP_000.pdf